CLINICAL TRIAL: NCT01056822
Title: Multicenter, Randomized, Open-label Study to Assess Whether Treatment With Mycophenolate Sodium (MPS) Allows Higher Dose Optimization Versus Mycophenolate Mofetil (MMF) Leading to a Dose Reduction of Tacrolimus. Maximiza Study.
Acronym: MAXIMIZA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080AES08; 2009-014562-26
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Prophilaxis of Acute Rejection in Patients Receiving a Renal Allograft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Mycophenolate mofetil
  Interventions: Drug: 1
- 2 (Experimental): Miycophenolate sodium
  Interventions: Drug: 2

INTERVENTIONS:
Drug: 1 — Continue with same dose of MMF as patient was taking before randomisation
  Arms: 1
Drug: 2 — Increase MPS by 180mg every 12h based on investigator's judgement up to a maximum of 720 mg of MPS every 12 hours
  Arms: 2

SUMMARY:
Multicenter, Randomized, Open-label Study to Assess Whether Treatment With Mycophenolate sodium (MPS) Allows Higher Dose Optimization Versus Mycophenolate mofetil (MMF) Leading to a Dose Reduction of Tacrolimus. Maximiza Study.

ELIGIBILITY:
Inclusion criteria

1. Renal transplant recipients ≥ 1 year and ≤ 5 years prior1 to inclusion in the study.
2. Patients who were receiving an immunosuppressive regimen including MMF ≤1000 mg/day and ≥ 250 mg/day 4 and Prograf®1 or Advagraf®6 (levels ≥7 ng/ml).
3. Patients who had been receiving the current maintenance immunosuppressive regimen with stable doses of MMF for at least the past 3 months.2
4. Patients included must have had Prograf® or Advagraf® levels ≥ 7ng/ml4 for at least one month prior to inclusion in the trial.2
5. Patients with low immunological risk, in the investigator's opinion.
6. Patients with an estimated glomerular filtration rate based on the MDRD formula of > 30 ml/min x 1.73 m2.1
7. Patients over 18 years of age.1
8. Patients who were able to understand the study information and give written informed consent.
9. Patients who were able to meet all study requirements, including completing questionnaires and attending study visits.

Exclusion criteria

1. Patients with GI symptoms known or assumed not to be caused by mycophenolic acid (MPA) treatment (e.g. oral bisphosphonate-induced infectious diarrhoea).
2. Patients with chronic inflammatory bowel disease.
3. Diabetic patients.
4. Acute rejection < 1 month prior to inclusion in the study.
5. Patients with leukopenia (< 3500 cells/mm3) or thrombocytopenia (< 100,000 cells/mm3).
6. Women of childbearing potential who were planning to become pregnant, were pregnant and/or breastfeeding, or who did not wish to use effective contraception [hormonal contraceptives (implantation, patches, oral) and double-barrier methods (any double combination of: IUD, male or female condoms with spermicidal gel, diaphragm, contraceptive sponge, cervical cap)].
7. Presence of psychiatric illness (such as schizophrenia, major depression) that, in the investigator's opinion, could interfere with study requirements.
8. Patients who were undergoing surgery for an acute condition or who were hospitalised.
9. Any other medical condition that, in the investigator's opinion based on blood counts or chart review, could interfere with completion of the study, including but not limited to visual problems or cognitive impairment.
10. Patients who were receiving or had received any investigational medicinal product during the 30 days prior to inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Spain (15):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Sodium (MPS): Participants continued their treatment with MPS according to normal clinical practice, with the dose of MPS increasing at each visit (visit 1 to visit 3) by 250 mg every 12 h and the dose of tacrolimus or tacrolimus extended release (ER) reducing by 25% (to a minimum level of 4 ng/ml).1 The purpose of dosage adjustments was to establish and maintain the patient on the maximum tolerated dose of MPS (up to a maximum of 1 g every 12 h).
- Mycophenolate Mofetil (MMF): Participants were converted to an equimolar dose of Mycophenolate mofetil at baseline visit. Dose of Mycophenolate mofetil was increased at each visit (visits 1 to visit 3) by 180 mg every 12 hours and the tacrolimus or tacrolimus extended release 6 dose was reduced by 25% (to a minimum level of 4 ng/ml). 1 Dosage adjustments allowed the patient to be established and maintained on the maximum tolerated dose of Mycophenolate mofetil (up to a maximum of 720 mg every 12 hours).
Period: Overall Study
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Started | 47 | 42
Intention-to-treat (ITT) Population: YES | 43 | 38
Intention-to-treat (ITT) Population: NO | 4 | 4
Per-protocol (PP) Population: YES | 29 | 25
Per-protocol (PP) Population: NO | 18 | 17
Safety (SAF) Population: YES | 46 | 40
Safety (SAF) Population: NO | 1 | 2
Completed | 39 | 35
Not Completed | 8 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 6 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population consisted of all randomised patients who gave signed informed consent and received at least one dose of the study medicinal product and have at least one baseline visit and one post-baseline visit (containing data to allow the primary endpoint to be calculated) Standard Deviation
Groups:
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF) | Total
Number analyzed (Participants) | 43 | 38 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.88 (9.99) | 48.50 (12.86) | 50.83 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 28 | 25 | 53
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 39 | 36 | 75
  Black | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Other | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving at Least Two Mycophenolic Acid (MPA) Dose Steps Higher and Reducing Tacrolimus Dose at the End of the Study
Time Frame: at 12 months from baseline
Population: Intention-to-treat (ITT) population included all randomised patients who gave signed informed consent and received at least one dose of study medicinal product and had at least one baseline visit and one post-baseline visit (containing data to allow primary endpoint to be calculated, i.e. dose of MPA or MMF and Tacrolimus).
Measure: Number; unit: number of participants
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 43 | 38
number of participants
  # of participants with ≥2 MPA dose steps higher | 0 | 0
  # of participants with <2 MPA dose steps higher | 43 | 38

2. Primary Outcome: Number of Participants That Achieved One Dose Step Higher With Mycophenolic Acid (MPA) or Mycophenolate Mofetil (MMF), According to the Treatment Group Assigned at the End of the Study (Final Visit) Compared to Baseline Dose
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Number; unit: study participants
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 43 | 38
study participants
  # of participants with ≥ 1 MPA dose steps higher | 37 | 30
  # of participants with < 1 MPA dose steps higher | 6 | 8

3. Primary Outcome: Participants With Reduction in Tacrolimus or Tacrolimus Extended Release Levels at the End of the Study (Final Visit) Compared to Baseline Dose.
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 43 | 38
Participants
  Reduction in tacrolimus or tacrolimus ER levels | 27 | 18
  No reduction in tacrolimus or tacrolimus ER levels | 16 | 20

4. Primary Outcome: Mean Mycophenolic Acid (MPA) Doses at the End of the Study (Final Visit) Compared to Baseline Dose.
Time Frame: at 12 months from baseline
Population: Per protocol (PP) population included all subjects from the ITT population who received medication throughout the study and did not have major protocol deviations and who participated in the study for a minimum of 210 days +/- 15 days
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 29 | 25
mg/day | 1173.10 (278.94) | 1195.20 (297.95)

5. Secondary Outcome: Change in Renal Function Measured Using Cockcroft-Gault Creatinine Clearance (CrCl)
Time Frame: Visit 1 (30 days +/-4), visit 2 (90 days +/- 15), visit 3 (150 days +/- 15), visit 4 (210 days +/- 15), visit 5 (365 days +/- 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/min
Units Other Than Participants: participants
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 43 | 38
ml/min
  Baseline (n=42,38) | 83.01 (26.51) | 83.44 (29.10)
  Visit 1 (n=41,37) | 81.55 (26.88) | 83.04 (27.06)
  Visit 2 (n=41,34) | 81.59 (26.60) | 82.88 (24.70)
  Visit 3 (n=37,35) | 84.91 (24.20) | 80.25 (23.25)
  Visit 4 (n=39,33) | 86.58 (26.82) | 81.83 (24.89)
  Visit 5 (n=36,33) | 88.08 (26.40) | 88.28 (29.17)

6. Secondary Outcome: Glomerular Filtration Rate (GFR) Using Abbreviated MDRD
Description: Calculated GFR (MDRD formula): GFR [mL/min/1.73m2] = 186.3*(C-1.154)*(A-0.203)*G*R where C is the serum concentration of creatinine [mg/dL], A is age [years], G=0.742 when gender is female, otherwise G=1, R=1.21 when race is black, otherwise R=1
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 43 | 38
mL/min/1.73m^2
  Baseline visit (n=43, 38) | 64.83 (17.59) | 61.08 (13.94)
  Visit 1 (n=42, 38; missings not included) | 62.68 (17.68) | 59.78 (12.32)
  Visit 2 (n=41, 35; missings not included) | 62.71 (17.02) | 60.84 (13.35)
  Visit 3 (n=40, 35; missings not included) | 67.74 (18.28) | 59.32 (13.71)
  Visit 4 (n=42, 36; missings not included) | 67.21 (20.19) | 61.20 (15.78)
  Visit 5 (n=38, 35; missings not included) | 70.24 (19.23) | 68.11 (19.84)

7. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS) Item Score
Description: The GSRS is a 15-item instrument design to assess the symptoms associated to gastrointestinal disorders. It has 5 subscales (reflux, diarrhoea, constipation, abdominal pain and indigestion) with scores rating from 1 to 7 (with a higher score representing more gastrointestinal symptoms)
Time Frame: as for outcome 5
Population: Intention-to-treat (ITT) population included all randomised patients who gave signed informed consent and received at least one dose of study medicinal product and had at least one baseline visit and one post-baseline visit (containing data to allow primary endpoint to be calculated, i.e. dose of MPA or MMF and Tacrolimus). Missings not included
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 43 | 38
Number analyzed (scores on a scale) | 43 | 38
scores on a scale
  Baseline Visit, Upper Abdomen Pain(n=42,37) | 1.64 (1.08) | 1.70 (1.02)
  Baseline Visit, Heartburn (n=42,37) | 1.29 (0.92) | 1.54 (1.41)
  Baseline visit, Acid reflux (n=42,37) | 1.40 (0.77) | 1.41 (0.98)
  Baseline visit, Hunger pains (n=43,37) | 2.30 (1.52) | 1.92 (1.21)
  Baseline visit, Nausea (n=43,37) | 1.30 (0.99) | 1.35 (0.95)
  Baseline visit, Rumbling in stomach (n=43,37) | 1.93 (1.12) | 1.92 (1.36)
  Baseline visit, Bloated (n=43,37) | 1.77 (1.27) | 2.27 (1.71)
  Baseline visit, Burping (n=43,37) | 1.91 (1.21) | 2.00 (1.39)
  Baseline visit, Passing gas/Flatus (n=43,37) | 2.19 (1.38) | 2.38 (1.48)
  Baseline visit, Constipation (n=42,37) | 1.71 (1.15) | 1.62 (1.36)
  Baseline visit, Diorrhoea (n=42,37) | 1.45 (1.09) | 1.51 (1.17)
  Baseline visit, Loose stool (n=42,37) | 1.69 (1.16) | 1.84 (1.38)
  Baseline visit, Hard stool (n=42,37) | 1.52 (1.04) | 1.65 (1.16)
  Baseline visit, Fecal incontinence (n=42,37) | 1.67 (1.18) | 2.03 (1.69)
  Baseline, Incomplete bowel emptying (n=42,37) | 1.57 (0.99) | 1.97 (1.36)
  Visit 2, Upper Abdomen Pain (n=40,34) | 1.43 (0.75) | 1.74 (1.16)
  Visit 2, Heartburn (n=40,35) | 1.43 (1.06) | 1.37 (0.73)
  Visit 2, Acid reflux (n=40,35) | 1.30 (0.76) | 1.57 (0.95)
  Visit 2, Hunger pains (n=39,34) | 2.33 (1.77) | 2.15 (1.33)
  Visit 2, Nausea (n=39,34) | 1.23 (0.67) | 1.29 (0.76)
  Visit 2, Rumbling in stomach (n=39,34) | 1.85 (1.06) | 1.85 (1.16)
  Visit 2, Bloated (n=40,35) | 1.73 (1.09) | 2.09 (1.48)
  Visit 2, Burping (n=40,35) | 1.80 (1.11) | 2.00 (1.55)
  Visit 2, Passing gas/Flatus (n=40,35) | 2.35 (1.42) | 2.34 (1.49)
  Visit 2, Constipation (n=40,33) | 1.58 (1.13) | 1.52 (0.97)
  Visit 2, Diorrhoea (n=40,33) | 1.38 (0.84) | 1.82 (1.42)
  Visit 2, Loose stool (n=40,32) | 1.73 (1.04) | 1.91 (1.20)
  Visit 2, Hard stool (n=39,35) | 1.51 (1.12) | 1.46 (0.82)
  Visit 2, Fecal incontinence (n=39,34) | 1.69 (1.30) | 2.12 (1.51)
  Visit 2, Incomplete bowel emptying (n=39,35) | 1.67 (0.96) | 1.69 (1.13)
  Visit 4, Upper Abdomen Pain (n=41,34) | 1.66 (1.26) | 2.00 (1.30)
  Visit 4, Heartburn (n=41,34) | 1.59 (1.24) | 1.74 (1.19)
  Visit 4, Acid reflux (n=41,34) | 1.46 (1.12) | 1.56 (0.99)
  Visit 4, Hunger pains (n=41,34) | 2.00 (1.60) | 2.26 (1.29)
  Visit 4, Nausea (n=41,34) | 1.37 (0.80) | 1.59 (1.18)
  Visit 4, Rumbling in stomach (n=41,34) | 2.02 (1.09) | 1.91 (1.22)
  Visit 4, Bloated (n=41,34) | 1.68 (1.04) | 2.15 (1.58)
  Visit 4, Burping (n=41,34) | 2.02 (1.41) | 2.21 (1.47)
  Visit 4, Passing gas/Flatus (n=41,34) | 2.46 (1.21) | 2.44 (1.48)
  Visit 4, Constipation (n=41,34) | 1.41 (0.74) | 1.85 (1.42)
  Visit 4, Diorrhoea ((n=41,34) | 1.59 (1.26) | 1.88 (1.09)
  Visit 4, Loose stool (n=41,34) | 2.00 (1.50) | 1.94 (1.13)
  Visit 4, Hard stool (n=40,34) | 1.53 (0.88) | 1.85 (1.26)
  Visit 4, Fecal incontinence (n=40,34) | 1.68 (1.29) | 2.12 (1.43)
  Visit 4, Incomplete bowel emptying(n=40,34) | 1.68 (0.92) | 1.88 (1.25)
  Visit 5, Upper Abdomen Pain (n=36,34) | 1.72 (1.19) | 1.85 (1.28)
  Visit 5, Heartburn (n=36,34) | 1.47 (0.94) | 1.56 (1.08)
  Visit 5, Acid reflux (n=36,34) | 1.25 (0.60) | 1.71 (1.14)
  Visit 5, Hunger pains (n=36,34) | 1.94 (1.49) | 2.12 (2.03)
  Visit 5, Nausea (n=36,34) | 1.28 (0.70) | 1.38 (0.92)
  Visit 5, Rumbling in stomach (n=36,34) | 2.03 (1.13) | 2.00 (1.41)
  Visit 5, Bloated (n=36,34) | 1.69 (1.12) | 2.12 (1.53)
  Visit 5, Burping (n=36,34) | 1.75 (1.18) | 2.00 (1.50)
  Visit 5, Passing gas/Flatus (n=36,34) | 2.33 (1.31) | 2.41 (1.60)
  Visit 5, Constipation (n=36,34) | 1.47 (0.91) | 1.68 (1.01)
  Visit 5, Diorrhoea (n=36,34) | 1.42 (1.02) | 1.71 (0.91)
  Visit 5, Loose stool (n=36,34) | 1.83 (1.23) | 1.74 (0.96)
  Visit 5, Hard stool (n=36,34) | 1.36 (0.72) | 1.79 (1.12)
  Visit 5, Fecal incontinence (n=36,34) | 1.86 (1.33) | 2.32 (1.70)
  Visit 5, Incomplete bowel emptying (n=36,34) | 1.69 (1.04) | 1.85 (1.18)

8. Secondary Outcome: Gastrointestinal Symptom Rating Scale (GSRS) Subscale Score
Description: as for outcome 7
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 43 | 38
Number analyzed (scores on a scale) | 43 | 38
scores on a scale
  Baseline visit, Indigestion (n=43,37) | 1.95 (0.89) | 2.14 (1.29)
  Baseline visit, Diorrhoea (n=41,37) | 1.58 (0.93) | 1.79 (1.26)
  Baseline visit, Constipation (n=41,37) | 1.59 (0.91) | 1.75 (1.12)
  Visit 2, Reflux (n=40,35) | 1.36 (0.81) | 1.47 (0.74)
  Visit 2, Abdominal pain (n=39,33) | 1.67 (0.71) | 1.71 (0.88)
  Visit 2, Indigestion (n=39,34) | 1.92 (0.87) | 1.96 (1.08)
  Visit 2, Diorrhoea (n=39,32) | 1.59 (0.94) | 1.94 (1.19)
  Visit 2, Constpation (n=39,33) | 1.59 (0.88) | 1.56 (0.86)
  Visit 4, Reflux (n=41,34) | 1.52 (1.15) | 1.65 (1.04)
  Visit 4, Abdominal pain (n=41,34) | 1.67 (0.83) | 1.95 (1.12)
  Visit 4, Indigestion (n=41,34) | 2.05 (0.97) | 2.18 (1.27)
  Visit 4, Diorrhoea (n=40,34) | 1.72 (1.23) | 1.98 (1.08)
  Visit 4, Constipation(n=40,34) | 1.54 (0.68) | 1.86 (1.12)
  Visit 5, Reflux (n=36,34) | 1.36 (0.69) | 1.63 (1.06)
  Visit 5, Abdominal pain (n=36,34) | 1.65 (0.66) | 1.78 (1.03)
  Visit 5, Indigestion (n=36,34) | 1.95 (0.95) | 2.13 (1.28)
  Visit 5, Diorrhoea (n=36,34) | 1.70 (1.02) | 1.92 (1.04)
  Visit 5, Constipation (n=36,34) | 1.51 (0.65) | 1.77 (0.89)

9. Secondary Outcome: Health-related Quality of Life (HRQoL): Impact of Gastrointestinal Symptoms on Quality Of Life (SIGIT)-QoL Questionnaire. Total Score.
Description: The SIGIT-QoL scale is a 17 items instrument, the score of each item ranges from 0 (always) to 4 (never). The scale score is obtained by adding the scores of the 17 items. Therefore, the total score ranges from 0 to 68 points. Higher score means, less impairment of Health Related QoL of the patient and vice versa, the lower the score, the greater severity of symptoms and worse perceived by the patient
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 43 | 38
Number analyzed (scores on a scale) | 43 | 38
scores on a scale
  Baseline visit (n=41,37) | 79.20 (6.86) | 76.00 (9.55)
  Visit 2 (n=38,32) | 78.79 (6.20) | 76.34 (10.12)
  Visit 4 (n=40,34) | 77.88 (6.64) | 74.53 (10.24)
  Visit 5, Diorrhoea (n=36,34) | 78.53 (5.06) | 76.41 (8.36)

10. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS) Score From Baseline to Visit 2 Stratified on the Basis of the Presence or Absence of Single-nucleotide Polymorphisms (SNPs) in the UGT1A9 Gene for the ITT Population
Description: Sub-study primary endpoint. The GSRS is a 15-item instrument design to assess the symptoms associated to gastrointestinal disorders. It has 5 subscales (reflux, diarrhoea, constipation, abdominal pain and indigestion) with scores rating from 1 to 7 (with a higher score representing more gastrointestinal symptoms)
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the UGT1A9 gene (n=3, 3) | 1.67 (10.50) | 0.00 (1.73)
  No SNP present in the UGT1A9 gene (n=18, 25) | -0.72 (6.52) | 1.52 (5.86)

11. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS) Score From Baseline to Visit 4 Stratified on the Basis of the Presence or Absence of Single-nucleotide Polymorphisms (SNPs) in the UGT1A9 Gene for the ITT Population
Description: as for outcome 10
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the UGT1A9 gene (n=4, 3) | 6.25 (12.39) | 0.67 (2.31)
  No SNP present in the UGT1A9 gene (n=19, 25) | 1.42 (9.06) | 2.96 (10.33)

12. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS) Score From Baseline to Visit 5 Stratified on the Basis of the Presence or Absence of Single-nucleotide Polymorphisms (SNPs) in the UGT1A9 Gene for the ITT Population
Description: as for outcome 10
Time Frame: at 12 months from baseline
Population: Intention-to-treat (ITT) population included all randomised patients who gave signed informed consent and received at least one dose of study medicinal product and had at least one baseline visit and one post-baseline visit (containing data to allow primary endpoint to be calculated, i.e. dose of MPA or MMF and Tacrolimus). Missing not included
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the UGT1A9 gene (n=3,3) | 8.00 (13.86) | 4.00 (4.00)
  No SNP present in the UGT1A9 gene (n=20, 23) | 1.10 (9.26) | -0.48 (9.55)

13. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS) Score From Baseline to Visit 2 Stratified on the Basis of the Presence or Absence of Single-nucleotide Polymorphisms (SNPs) in the MRP2 Gene for the ITT Population
Description: as for outcome 10
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the MRP2 gene (n=9, 14) | 1.78 (6.65) | 0.79 (5.91)
  No SNP present in the MRP2 gene (n=12, 14) | -2.00 (6.94) | 1.93 (5.36)

14. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS) Score From Baseline to Visit 4 Stratified on the Basis of the Presence or Absence of Single-nucleotide Polymorphisms (SNPs) in the MRP2 Gene for the ITT Population
Description: as for outcome 10
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the MRP2 gene (n=9, 14) | 5.67 (11.48) | 3.71 (6.23)
  No SNP present in the MRP2 gene (n=14, 14) | 0.07 (7.79) | 1.71 (12.57)

15. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS) Score From Baseline to Visit 5 Stratified on the Basis of the Presence or Absence of Single-nucleotide Polymorphisms (SNPs) in the MRP2 Gene for the ITT Population
Description: as for outcome 10
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the MRP2 gene (n=9, 14) | 3.67 (10.17) | 1.92 (9.40)
  No SNP present in the MRP2 gene (n=14, 14) | 0.93 (9.88) | -1.57 (8.94)

16. Secondary Outcome: Change in SIGIT-QoL Score From Baseline to Visit 2 Stratified on the Basis of the Presence or Absence of SNP in the UGT1A9 Gene for the ITT Population
Description: Sub-study primary endpoint. The SIGIT-QoL scale is a 17 items instrument, the score of each item ranges from 0 (always) to 4 (never). The scale score is obtained by adding the scores of the 17 items. Therefore, the total score ranges from 0 to 68 points. Higher score means, less impairment of Health Related QoL of the patient and vice versa, the lower the score, the greater severity of symptoms and worse perceived by the patient
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the UGT1A9 gene (n=4, 3) | -5.50 (6.45) | 0.33 (0.58)
  No SNP present in the MRP2 gene (n=18, 28) | -0.44 (2.81) | -0.46 (5.35)

17. Secondary Outcome: Change in SIGIT-QoL Score From Baseline to Visit 4 Stratified on the Basis of the Presence or Absence of SNP in the UGT1A9 Gene for the ITT Population
Description: as for outcome 16
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the UGT1A9 gene (n=4, 3) | -5.75 (7.41) | -1.67 (2.52)
  No SNP present in the UGT1A9 gene (n=19, 27) | -2.00 (7.14) | -2.63 (8.54)

18. Secondary Outcome: Change in SIGIT-QoL Score From Baseline to Visit 5 Stratified on the Basis of the Presence or Absence of SNP in the UGT1A9 Gene for the ITT Population
Description: as for outcome 16
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the UGT1A9 gene (n=3, 3) | -1.33 (8.39) | -3.67 (6.35)
  No SNP present in the UGT1A9 gene (n=20, 26) | -0.55 (5.45) | -0.65 (7.03)

19. Secondary Outcome: Change in SIGIT-QoL Score From Baseline to Visit 2 Stratified on the Basis of the Presence or Absence of SNP in the MRP2 Gene for the ITT Population
Description: Sub-study primary endpoint. SIGIT-QoL scale is a 17 items instrument, the score of each item ranges from 0 (always) to 4 (never). The scale score is obtained by adding the scores of the 17 items. Therefore, the total score ranges from 0 to 68 points. Higher score means, less impairment of Health Related QoL of the patient and vice versa, the lower the score, the greater severity of symptoms and worse perceived by the patient
Time Frame: at 12 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the MRP2 gene (n=9,16) | -0.89 (3.79) | 0.56 (4.65)
  No SNP present in the MRP2 gene (n=13, 15) | -1.69 (4.33) | -1.40 (5.49)

20. Secondary Outcome: Change in SIGIT-QoL Score From Baseline to Visit 4 Stratified on the Basis of the Presence or Absence of SNP in the MRP2 Gene for the ITT Population
Description: as for outcome 16
Time Frame: at 12 months from baseline
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the MRP2 gene (n=9,15) | -2.67 (7.78) | -1.73 (5.40)
  No SNP present in the MRP2 gene (n=14, 15) | -2.64 (7.04) | -3.33 (10.29)

21. Secondary Outcome: Change in SIGIT-QoL Score From Baseline to Visit 5 Stratified on the Basis of the Presence or Absence of SNP in the MRP2 Gene for the ITT Population
Description: as for outcome 16
Time Frame: at 12 months from baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: scores on a scale
Arm/Group | Mycophenolate Sodium (MPS) | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 24 | 31
Number analyzed (scores on a scale) | 24 | 31
scores on a scale
  SNP present in the MRP2 gene (n=9,14) | -1.11 (6.86) | -0.50 (7.85)
  No SNP present in the MRP2 gene (n=14, 15) | -0.36 (5.02) | -1.40 (6.17)

22. Secondary Outcome: Duration of Exposure to the Study Medicinal Product, Mycophenolate Sodium Descriptive Statistics. Safety Population Per Treatment Group
Description: Exposure to study drug (MPS). Data presented only for safety population on the study treatment arm (not applicable for MMF arm)
Time Frame: at 12 months from baseline
Population: The safety population included all randomised patients who gave signed informed consent and received at least one dose of the study medicinal product.
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: participants
Arm/Group | Mycophenolate Sodium (MPS)
Number analyzed (Participants) | 46
days | 201.91 (49.00)

23. Secondary Outcome: Dose of the Study Medicinal Product Mycophenolate Sodium (MPS)
Description: Safety population per visit and per treatment group
Time Frame: at 12 months from baseline
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Units Other Than Participants: patient doses
Arm/Group | Mycophenolate Sodium (MPS)
Number analyzed (Participants) | 46
Number analyzed (patient doses) | 46
mg
  Baseline visit (n=46) | 579.13 (165.03)
  Visit 1 (n=43) | 856.28 (181.65)
  Visit 2 (n=41) | 1080.00 (238.12)
  Visit 3 (n=40) | 1228.50 (263.81)

24. Secondary Outcome: Dose of the Study Medicinal Product Mycophenolate Mofetil (MMF)
Description: Safety population per visit and per treatment group (missings not included)
Time Frame: at 12 months from baseline
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg
Units Other Than Participants: patient doses
Arm/Group | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 40
Number analyzed (patient doses) | 40
mg
  Baseline visit (n=40) | 806.25 (222.80)
  Visit 1 (n=38) | 1250.00 (278.75)
  Visit 2 (n=35) | 1578.57 (382.39)
  Visit 3 (n=35) | 1757.14 (381.01)

ADVERSE EVENTS:
Groups:
- Micofenolato Sodium: Micofenolato sodium
- Micofenolato Mofetilo: Micofenolato mofetilo
Arm/Group | Micofenolato Sodium | Micofenolato Mofetilo
Serious Adverse Events (participants affected / at risk) | 2/46 | 4/40
Other Adverse Events (participants affected / at risk) | 13/46 | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micofenolato Sodium (N=46) | Micofenolato Mofetilo (N=40)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 0 | 1
Human polyomavirus infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Micofenolato Sodium (N=46) | Micofenolato Mofetilo (N=40)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 1 | 2
Urinary tract infection (Infections and infestations) | 5 | 1
Blood creatinine increased (Investigations) | 1 | 2
Headache (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or disclosure of the trial results in their entirety.